CLINICAL TRIAL: NCT05178745
Title: A Prospective Observational Cohort Study Evaluating Resection Rate in Patients With Metastatic Colorectal Cancer Treated With Aflibercept in Combination With FOLFIRI - Observatoire résection
Brief Title: Resection Observatory
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS15624; AFLIBL07747 (Other: Sanofi); U1111-1272-2417 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Colorectal Cancer; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; aflibercept; Irinotecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with metastatic colorectal cancer and liver metastases treated with FOLFIRI plus aflibercept after failure of an oxaliplatin-based regimen
  Interventions: Drug: Fluorouracil; Drug: Aflibercept; Drug: Irinotecan

INTERVENTIONS:
Drug: Fluorouracil — Pharmaceutical Form: solution for injection Route of Administration: intravenous (IV), intravenous or intra-arterial infusion
Drug: Aflibercept — Pharmaceutical Form: concentrate solution for infusion Route of Administration: IV infusion
  Other Names: ZALTRAP®
Drug: Irinotecan — Pharmaceutical Form: solution for injection Route of Administration: IV infusion
  Other Names: CAMPTOSAR®

SUMMARY:
Primary Objective:

-Evaluate the resection rate (R0/R1) in current practice for aflibercept in combination with irinotecan plus 5-fluorouracil (FOLFIRI) in patients treated for metastatic colorectal cancer (mCRC) after failure of an oxaliplatin-containing regimen

Secondary Objectives:

* Evaluate overall survival, progression-free survival and relapse-free survival.
* Evaluate conversion rates (initially unresectable disease which became resectable after chemotherapy, with R0/R1 resection).
* Evaluate histological and radiological response rates.
* Evaluate rate of postoperative complications.
* Evaluate safety.

DETAILED DESCRIPTION:
The estimated inclusion period is 45 months. Patient follow-up is 24 months and the total study duration is 69 months. Last patient status (alive or dead) collected before database lock.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with aflibercept in combination with FOLFIRI for mCRC after failure of an oxaliplatin-containing regimen (including patients pretreated with bevacizumab or anti-EGFR and patients treated with oxaliplatin in the adjuvant setting).
* Exclusively or predominantly hepatic metastases (≤ 5 pulmonary nodules < 2 cm).
* Age > 18 years.
* Signed consent for collection of personal and medical data.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.

Exclusion Criteria:

* Concomitant participation in a clinical trial.
* Patient receiving concomitant anti-VEGF agents and/or receiving aflibercept as part of a clinical trial or in a compassionate use program.
* Patient receiving aflibercept in combination with chemotherapy other than FOLFIRI.
* Patient with contra-indication to surgery.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this study will be patients treated with aflibercept in combination with FOLFIRI for metastatic ColoRectal Cancer (mCRC) after failure of an oxaliplatin-containing regimen (including patients pretreated with bevacizumab or anti-estimated glomerular filtration rate (anti-EGFR) and patients treated with oxaliplatin in the adjuvant setting but excluding these already participating in a clinical trial) recruited from particpating sites in France. The study will aim to enroll approximately 140 adult patients treated with aflibercept in combination with FOLFIRI for metastatic colorectal cancer after failure of an oxaliplatin-containing regimen from up to 30 sites.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Assessment of resection rate (R0/R1) | Up to 24 months
  R0 /R1 resection rate after aflibercept + FOLFIRI (resection with histological assessment of margin status)

SECONDARY OUTCOMES:
Overall survival | Up to 69 months
  Defined starting from the date of the first aflibercept administration.
Progression-free surivival | Up to 69 months
  Defined as the time from the date of the first aflibercept administration to the date of the first event (progression, relapse or death). (Relapse in case of complete response due to chemotherapy or surgery)
Relapse-free surivial | Up to 69 months
  Defined as the time from the date of the first aflibercept administration to the date of the first event (progression, relapse or death). (Relapse in case of complete response due to chemotherapy or surgery)
Objective Response | Up to 69 months
  Assessed according to RECIST and CHUN (radiological assessment) criteria in the exploratory analysis.
Conversion rate | Up to 69 months
  Initially unresectable disease which became resectable after aflibercept + FOLFIRI, with R0/R1 resection).
Histological response of resected patients via Tumor Regression Grade (TRG) | Up to 69 months
  Histological response of resected patients via TRG
Histological response of resected patients via Modified Tumor Regression Grade (mTRG) | Up to 69 months
  Histological response of resected patients via mTRG,
Histoligical response of resected patients via Blazer assessment | Up to 69 months
Histological response of resected patients via modified Blazer assessment | Up to 69 months
Histological response of resected patients via Sebagh assessment | Up to 69 months
Radiological response for all patients using RECIST 1.1 criteria | Up to 69 months
Rate of 90-day postoperative complications using DINDO-CLAVIEN classification | Up to 69 months
Safety (serious and non-serious adverse events occurring during treatment | Up to 69 months
  Number of patients with serious and non-serious adverse events occurring during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Tougeron D, Bibeau F, Chibaudel B, Kim S, Nguyen T, Phelip JM, Mille D, Bouattour M, Tavan D, Rinaldi Y, Lecomte T, Perrier H, Spaeth D, Caroli Bosc FX, Metges JP, Ferec M, Hautefeuille V, Deslandres-Cruchant M, Danion J, Hammel P, Lewin M, Tasu JP, Angelergues A, DiFiore F, Evrard S, Mansar R, Caillou H, Geffriaud-Ricouard C, Adam R. Resection of colorectal liver metastases with second-line aflibercept plus FOLFIRI: Results from the RESECTION prospective French cohort. Eur J Cancer. 2024 Dec;213:115082. doi: 10.1016/j.ejca.2024.115082. Epub 2024 Oct 22. PMID 39486163